CLINICAL TRIAL: NCT03350529
Title: Feasibility and Safety of Transurethral HIFU in Various Prostate Diseases; Particularly Prostate Cancer
Brief Title: MRI Guided Transurethral HIFU for Various Prostate Diseases
Acronym: HIFU-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TO3/001/17
Record Dates: First submitted 2017-10-12; First posted 2017-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Localised Prostate Cancer; Locally Advanced Prostate Cancer; Locally Recurrent Prostate Cancer; Benign Prostatic Hyperplasia
Keywords: prostate cancer; benign prostatic hyperplasia; benign prostatic obstruction; high intensity focused ultrasound; real-time temperature feedback control; magnetic resonance imaging
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is an early phase 1 non-randomized prospective single-institutional and four arm study to determine the applicability, feasibility and safety of MRI guided transurethral HIFU ablation of prostate separately in each pre-specified group/arm (10 patients per group).
  Due to the encouraging feasibility and safety results, an amendment was made to the original study protocol to increase the amount of salvage group patients and BPH group patients. With the approval of the ethics committee, the sample size of the salvage group and BPH group was increased to a total of 40 patients and 30 patients, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Localised PC prior to RP (Experimental): MRI guided transurethral HIFU ablation is targeted to MRI visible, biopsy proven, index lesion(s) within prostate and if possible with 5mm angular extension (imaging based healthy tissue marginal) to both sides from the tumour boundary in transverse plane and 5 mm in coronal plane. The ablative effect is aimed to reach prostate capsule by heating the control boundary (3 mm from capsule) to temperature 57 °C. The focal approach is intended to be radical as for index lesion.
  Interventions: Device: MRI guided transurethral HIFU ablation of prostatic tissue
- Symptomatic locally advanced PC (Experimental): MRI guided transurethral HIFU ablation is targeted to main prostatic malignant tumour squeezing and/or invading the prostatic urethra and/or bladder neck. The approach is intended to be palliative.
  Interventions: Device: MRI guided transurethral HIFU ablation of prostatic tissue
- Locally recurrent PC after EBRT (Experimental): MRI guided transurethral HIFU ablation is targeted to MRI visible, biopsy proven, local recurrent index lesion(s) within and/or surrounding prostate and if possible with 5 mm angular extension to either side from the tumour boundary in transverse plane and 5 mm in coronal plane. The approach is intended to be focal and salvage.
  The whole-gland HIFU ablation approach will be considered in case of extensive organ confined recurrent prostate cancer (positive biopsies for malignancy from extensive/multiple area in prostate and/or extensive/multiple lesion(s) at baseline MRI) to cover whole prostate.
  Interventions: Device: MRI guided transurethral HIFU ablation of prostatic tissue
- Symptomatic BPH (Experimental): MRI guided transurethral HIFU ablation is targeted to adenomas of the prostate. The HIFU sector encompasses bilateral (anterolateral) transitional zones between bladder neck and verumontanum (colliculus seminalis).
  Interventions: Device: MRI guided transurethral HIFU ablation of prostatic tissue

INTERVENTIONS:
Device: MRI guided transurethral HIFU ablation of prostatic tissue — The technology is developed to ablate targeted benign and malignant prostate tissue through transurethrally inserted probe that transmit ultrasound energy under MRI guidance and control. The therapeutic endpoint of this method is thermal coagulation of prostate tissue.
  Other Names: TULSA-PRO (Profound Medical Inc), Device: PAD-105

SUMMARY:
This study assesses feasibility and safety, the primary outcomes, of MRI guided transurethral high intensity focused ultrasound (HIFU) ablation for prostate diseases (PD). We will enrol 10 patients to each group with criteria as follows: localised prostate cancer (PC); locally advanced PC; locally recurrent PC after external beam radiation therapy (EBRT); benign prostatic hyperplasia (BPH). Secondary outcomes are both oncologic and functional outcomes and imaging based follow up after HIFU therapy will be also assessed.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common cancer among men in Finland with the highest incidence of all cancers. Benign prostate hyperplasia (BPH) also has high prevalence, increasing with age. BPH may cause harmful lower urinary tract symptoms (LUTS) and it is demonstrated that by the age of 60, over 50 % of men have clinically significant prostate BPH and up to 40 % of men over age 60 suffer from LUTS.

Currently curative intended therapies for PC, radiation therapy (RT) and radical prostatectomy (RP), offer desirable oncologic local control but have major impact on genitourinary function and quality of life (QoL). Some patients are unfit for surgical procedures or cannot tolerate RT due to concomitant medical conditions or prior therapies. At present lower risk PC is increasingly managed with active surveillance. However, diagnosis of PC and active surveillance itself may both lead to notable psychological and emotional burden impairing QoL. Further, significant amount of cases in some point end up in radical treatment resulted from either risk profile upgrade or patients preference. For these patients optimal treatment might be a focal therapy with sufficient oncologic control and minor impact on QoL.

There is controversy related to optimal treatment in local recurrence after RT. 45% of patients will have local recurrence after RT within 8 years after treatment. Androgen deprivation therapy (ADT) decelerate disease only temporarily and salvage RP includes major risks and is technically demanding, but can provide long-term cure in selected patients.

On the aspect of palliation, there is an eminent need for less invasive supplementary therapies since patients presenting with metastatic or locally advanced PC, generally have low performance status.

Management of benign prostatic obstruction has also faced challenges with conventional treatment modalities, since ageing and profuse co-morbidities among patients have increased. Transurethral resection of prostate (TURP) is still the standard treatment in severe LUTS caused by BPH.

Recently the major development of magnetic resonance imaging (MRI) has been achieved improving PC diagnosis and local staging. Even though PC is often multifocal, evidence indicates that both clinical outcome and prognosis of PC is determined predominantly by index lesion. Because of the notable risk of morbidities involving radical treatments and significant evolution of MRI, focal therapies have attained wide interest. One of the most interesting focal mini-invasive treatment is high intensity focused ultrasound (HIFU). HIFU technique exploits thermal energy; by raising target temperature over 55°C target volume is destroyed due to acute coagulation necrosis. Modern devices delivering HIFU to the prostate are transurethral and emit directional high intensity ultrasound to the focused regions utilising superior MRI guidance compared to older generation ultrasound guidance. Magnetic resonance thermometry technique utilizes noninvasive measurement of tissue temperature allowing monitoring real time temperature changes during treatment. The MRI treatment system is equipped with active dynamic temperature feedback control designed to maintain a constant temperature inside the target volume and at the boundary of the target area. By this way conformal three-dimensional ablative volumes with great spatial accuracy and precision can be achieved simultaneously avoiding damages to the surrounding sensitive tissues. Therapy verification is confirmed instantaneously after treatment by acquiring contrast enhanced MRI (CE-MRI) that visualise the non-perfused-volume (NPV) describing the success of total ablation of the target prostate volume.

This prospective clinical single center feasibility and safety study will evaluate the role of MRI guided transurethral HIFU ablation for various PD and clinical settings. All enrolled patients have prostate pathology and different clinical situation with need of definitive interventions and they are divided to four arms/groups according to specific inclusion criterion. Group 1 localised PC prior to RP, group 2 symptomatic locally advanced PC in need of palliative surgical intervention, group 3 locally recurrent PC after EBRT and group 4 symptomatic BPH in need for intervention.

The hypothesis is that MRI guided transurethral HIFU is feasible and safe in various prostate diseases and clinical settings. If hypothesis is proven for certain or for all groups, the investigators will continue with that group or groups to phase 2 clinical multi-institutional studies.

ELIGIBILITY:
Shared inclusion criteria for all groups:

* Language spoken: Finnish, English or Swedish
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff.
* Potential prostate biopsies obtained > 6 weeks before HIFU/TULSA-PRO treatment (or at the discretion of PI)
* Eligible for MRI
* Eligible for spinal or general anesthesia (ASA 3 or less)
* Succession of urethral catheterization/Patency of prostatic urethra confirmed if needed with pre-HIFU cystoscopy

Group-specific inclusion criteria

Group 1. Localized PC prior to RP

* All localized PC patients planned for robot assisted laparoscopic prostatectomy (RALP) with normal standards of care are eligible for this study (EAU guidelines)
* MRI-visible biopsy proven PC (biopsies obtained < 6 months before treatment)

Group 2. Locally symptomatic locally advanced and/or metastatic prostate cancer in need of palliative surgical intervention

* gross recurrent hematuria
* bladder outlet obstruction with intractable symptoms
* urinary retention

Group 3. Locally recurrent PC after EBRT as a salvage approach

* Phoenix criteria of biochemical relapse (PSA nadir + 2 ng/ml)
* MRI-visible, biopsy proven local recurrence
* No evidence of distant metastasis in PSMA-PET/CT

Group 4. Symptomatic BPH with need for intervention

* Patients planned for surgical procedure (e.g. TURP, laservaporization or open adenomectomy) with normal standards of care are eligible for this study
* Bilobular hyperplasia (enlarged transition zone lobes) without dominant enlargement of periurethral zone "median lobe" assessed in cystoscopy and TRUS
* No suspicion of cancer on baseline MRI (PI-RADS v2 lesion < 3)

Shared exclusion criteria for all groups:

* Prostate calcifications >1cm in largest diameter located in the anticipated treatment sector on baseline TRUS or MRI
* Prostate cysts >1cm in largest diameter located in the anticipated treatment sector on baseline TRUS or MRI
* History of chronic inflammatory conditions (e.g. inflammatory bowel disease) affecting rectum (also includes rectal fistula and anal/rectal stenosis)
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc.)
* Uncontrolled serious infection
* Claustrophobia
* Hip replacement surgery or other metal in the pelvic area
* Severe kidney failure (glomerular filtration rate (GFR) <30ml/min/1.73m2) exclude usage of gadolinium in contrast-enhanced imaging unless justifiable based on the clinical judgment of the responsible radiologist and/or urologist.
* Known allergy to gadolinium
* Known allergy or contraindication to GI anti-spasmodic drug (e.g. glucagon, buscopan)
* Inability to insert urinary catheter (i.e. urethral stricture disease)
* Patients with artificial urinary sphincter, urethral sling or any penile implant
* Any other conditions that might compromise patient safety, based on the clinical judgment of the responsible urologist

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate targeting accuracy of HIFU ablation separately in each study arm/group. | The date of HIFU treatment
  Quantitative analysis of targeting accuracy is defined as spatial difference between target prostate region in treatment planning phase and the target temperature isotherm (57°C) at the end of HIFU treatment on MRI thermometry. The measure used is dice similarity coefficient (DSC - unitless from 0 to 1) which is a statistical validation metric to measure the degree of spatial overlap between two regions.
  The measure is a composite outcome measure reported as single value for each arm/group.
Evaluate targeting accuracy volume of HIFU ablation separately in each study arm/group. | The date of HIFU treatment
  Quantitative analysis of targeting accuracy volume illustrates over- and under-treatment representing the amount of tissue ≥ target temperature 57°C outside the target volume and < target temperature 57°C inside the target volume, respectively.
  Over- and under-treatment volumes are expressed as a % of the target volume.
  The measure is a composite outcome measure reported as single value for each arm/group.
Radiologically determined treatment accuracy of HIFU ablation in localised PC arm/group. | 3-4 weeks from the treatment date
  Quantitative analysis of radiologically verified treatment accuracy; determined by comparing targeting volumes on MRI during treatment planning to immediate, 1 and 3 week NPV in CE-MRI following HIFU therapy. The ratio in percentage (%) between target prostate volume (ml) and NPV (ml) will be measured.
Histopathologically determined treatment accuracy of HIFU ablation in localised PC arm/group. | 3-4 weeks from the treatment date
  Qualitative analysis of treatment accuracy; determined by comparing both targeting volume on MRI during treatment planning and immediate, 1 and 3 weeks NPV following HIFU therapy separately to histopathologically verified coagulation necrosis volume from the removed prostate at 3 week after HIFU therapy. The ratio in percentage between target prostate volume (ml) and NPV (ml) to coagulative necrosis volume (ml) will be measured.
Radiologically determined treatment accuracy of HIFU ablation in locally advanced PC arm/group. | 12 months from the treatment date
  Quantitative analysis of treatment accuracy; determined by comparing targeting volume on MRI during treatment planning to immediate, 1 week and 12 months NPV in CE-MRI following HIFU therapy.
  The ratio in percentage between target prostate volume (ml) and NPV (ml) will be measured.
Radiologically determined treatment accuracy of HIFU ablation in locally recurrent PC after EBRT arm/group. | 12 months from the treatment date
  Quantitative analysis of treatment accuracy; determined by comparing targeting volume on MRI during treatment planning to immediate, 1 week and 12 months NPV in CE-MRI following HIFU therapy.
  The ratio in percentage between target prostate volume (ml) and non-perfused volume (ml) will be measured.
Radiologically determined treatment accuracy of HIFU ablation in BPH arm/group. | 12 months from the treatment date
  Quantitative analysis of treatment accuracy; determined by comparing targeting volume on MRI during treatment planning to immediate, 1 week and 12 months NPV in CE-MRI following HIFU therapy. The ratio in percentage between target prostate volume (ml) and NPV (ml) will be measured.
Safety of MRI guided transurethral HIFU ablation in various prostate diseases | 12 months from the treatment date
  Safety is determined in each group and all group together by evaluation of the frequency and severity of device/treatment related adverse events associated with the use of TULSA-PRO system to ablate prostate tissue. The severity of the adverse events are graded according to the Clavien-Dindo Classification of surgical complications.
  The measure is a composite outcome measure reported as single value for each arm/group.

SECONDARY OUTCOMES:
Preliminary efficacy of HIFU ablation to achieve sufficient tumour control in patients having local recurrent PC after EBRT | 12 months from the treatment date
  Histopathological evaluation of the treatment response is based on 2-6-core biopsy results obtained from HIFU treated region/volume at 12 months. The number of biopsies taken is depended on the size and extension of the primary lesion treated with HIFU. The cognitive transrectal ultrasound guided biopsy method will be used to confirm histologically anticipated treatment success; coagulative necrosis/fibrosis/scar tissue of the prostate tissue. The outcome of biopsies (negativity/positivity for prostate cancer) will be measured. The proportion of patients with negative prostate biopsy will be measured at 12 months follow-up visit.
Image based follow up following HIFU ablation | 12 months from the treatment date
  Evaluation and characterisation of image based follow up with repetitive mpMRI (Arm/group 1: immediate, 1 and 3 week, Arms/Groups 2, 3 and 4: immediate, 1 week, 12 month) after HIFU treatment. Image based follow up will be focused on modifications and development of the rim of enhancement surrounding NPV and the evolution of NPV following HIFU treatment.

OTHER OUTCOMES:
Preliminary efficacy of MRI guided transurethral HIFU ablation in locally recurrent PC after EBRT in terms of serum PSA response. | 12 months from the treatment date
  Explore and characterise short- and medium-term pattern of S-PSA response following HIFU ablation. Serum PSA will be measured before HIFU ablation and predetermined interval during follow up protocol after HIFU ablation. The serum PSA trend and nadir following HIFU ablation will be demonstrated.
Evaluate voiding function by using uroflowmetry before and after HIFU ablation separately in each arm/group. | 12 months from the treatment date
  Voiding function is assessed separately in each group/arm by:
  - measuring the rate of flow of voided urine using a flowmeter, a device that measures the quantity of urine (volume) voided per unit time (uroflowmetry). The measurement is expressed in millilitres per second (ml/s).
  The data from uroflowmetry before and after HIFU ablation will be compared.
Evaluate voiding function by measuring PVR before and after HIFU ablation separately in each arm/group. | 12 months from the treatment date
  Voiding function is assessed separately in each group/arm by:
  - post-voided residual urine (PVR) (volume in ml), which estimates the completeness of bladder emptying using a handheld ultrasonic bladder scanner.
  The PVR before and after HIFU ablation will be compared.
Evaluation of QoL following HIFU ablation in each prostate cancer arm/group | 12 months from the treatment date
  Evaluation of QoL using standardised questionnaire:
  - 26-item short-form version of EPIC, The Expanded Prostate Index Composite
  QoL questionnaire before and after HIFU ablation are compared.
  The measure is a composite outcome measure reported as single value for each arm/group.
Evaluation of change in urinary symptoms following HIFU ablation in BPH group | 12 months from the treatment date
  Quality of life questionnaire, International Prostate Symptom Score (IPSS), is used to assess urinary symptoms following HIFU therapy. IPSS consists of seven question concerning urinary symptoms (points from 0 to 5) and one separate question concerning quality of life (points from 0 to 6). The total score of questions related to urinary symptoms can range from 0 to 35. The baseline IPSS score is compared to IPSS scores obtained from predetermined follow up protocol following HIFU therapy to characterise HIFU therapy´s short- (1 week, 3 and 6 months) and medium-term (12 months) impact on lower urinary tract function. A significant change in IPSS is defined as a change of > 3 points.
  The change in total points of IPSS between baseline and most recent follow up visit is measured.
Evaluation of change in erectile function following HIFU ablation in BPH group | 12 months from the treatment date
  Quality of life questionnaire, International Index of Erectile Function (IIEF-15), is used to assess sexual function following HIFU therapy. A score of 0-5 is awarded to each of the 15 questions that examine 4 main domain of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  Change in total score and each domain of IIEF-15 separately are measured between the baseline and most recent follow-up visit.
Evaluate painfulness of HIFU therapy in treating various prostate diseases | 12 months from the treatment date
  The pain is assessed predetermined interval during follow up using Visual Analog Scale for pain (VAS for pain, numerical rating scale 1-10).
  The measure is a composite outcome measure reported as single value for each arm/group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, M.D.Ph.D, Principal Investigator — Department of Urology, VSSHP, University of Turku
Locations (1):
- Department of Urology, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.www.cancerregistry.fi
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Wasserman NF. Benign prostatic hyperplasia: a review and ultrasound classification. Radiol Clin North Am. 2006 Sep;44(5):689-710, viii. doi: 10.1016/j.rcl.2006.07.005. PMID 17030221
- [Background] 4. McDougal WS, Wein AJ, Kavoussi LR, et al: Campbell-Walsh Urology 10th Edition Review E-Book. A Saunders Title; 2011. p. 704
- [Background] McNeal JE. Anatomy of the prostate and morphogenesis of BPH. Prog Clin Biol Res. 1984;145:27-53. No abstract available. PMID 6201879
- [Background] Cooperberg MR, Moul JW, Carroll PR. The changing face of prostate cancer. J Clin Oncol. 2005 Nov 10;23(32):8146-51. doi: 10.1200/JCO.2005.02.9751. PMID 16278465
- [Background] Bechis SK, Carroll PR, Cooperberg MR. Impact of age at diagnosis on prostate cancer treatment and survival. J Clin Oncol. 2011 Jan 10;29(2):235-41. doi: 10.1200/JCO.2010.30.2075. Epub 2010 Dec 6. PMID 21135285
- [Background] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Background] Potosky AL, Davis WW, Hoffman RM, Stanford JL, Stephenson RA, Penson DF, Harlan LC. Five-year outcomes after prostatectomy or radiotherapy for prostate cancer: the prostate cancer outcomes study. J Natl Cancer Inst. 2004 Sep 15;96(18):1358-67. doi: 10.1093/jnci/djh259. PMID 15367568
- [Background] van Tol-Geerdink JJ, Leer JW, van Oort IM, van Lin EJ, Weijerman PC, Vergunst H, Witjes JA, Stalmeier PF. Quality of life after prostate cancer treatments in patients comparable at baseline. Br J Cancer. 2013 May 14;108(9):1784-9. doi: 10.1038/bjc.2013.181. Epub 2013 Apr 23. PMID 23612450
- [Background] Klotz L. Expectant management with selective delayed intervention for favorable risk prostate cancer. Urol Oncol. 2002 Sep-Oct;7(5):175-9. doi: 10.1016/s1078-1439(02)00183-7. PMID 12644212
- [Background] Reeve BB, Stover AM, Jensen RE, Chen RC, Taylor KL, Clauser SB, Collins SP, Potosky AL. Impact of diagnosis and treatment of clinically localized prostate cancer on health-related quality of life for older Americans: a population-based study. Cancer. 2012 Nov 15;118(22):5679-87. doi: 10.1002/cncr.27578. Epub 2012 Apr 27. PMID 22544633
- [Background] Bul M, Zhu X, Valdagni R, Pickles T, Kakehi Y, Rannikko A, Bjartell A, van der Schoot DK, Cornel EB, Conti GN, Boeve ER, Staerman F, Vis-Maters JJ, Vergunst H, Jaspars JJ, Strolin P, van Muilekom E, Schroder FH, Bangma CH, Roobol MJ. Active surveillance for low-risk prostate cancer worldwide: the PRIAS study. Eur Urol. 2013 Apr;63(4):597-603. doi: 10.1016/j.eururo.2012.11.005. Epub 2012 Nov 12. PMID 23159452
- [Background] Nguyen PL, D'Amico AV, Lee AK, Suh WW. Patient selection, cancer control, and complications after salvage local therapy for postradiation prostate-specific antigen failure: a systematic review of the literature. Cancer. 2007 Oct 1;110(7):1417-28. doi: 10.1002/cncr.22941. PMID 17694553
- [Background] Kuban DA, Thames HD, Levy LB, Horwitz EM, Kupelian PA, Martinez AA, Michalski JM, Pisansky TM, Sandler HM, Shipley WU, Zelefsky MJ, Zietman AL. Long-term multi-institutional analysis of stage T1-T2 prostate cancer treated with radiotherapy in the PSA era. Int J Radiat Oncol Biol Phys. 2003 Nov 15;57(4):915-28. doi: 10.1016/s0360-3016(03)00632-1. PMID 14575822
- [Background] Heidenreich A, Richter S, Thuer D, Pfister D. Prognostic parameters, complications, and oncologic and functional outcome of salvage radical prostatectomy for locally recurrent prostate cancer after 21st-century radiotherapy. Eur Urol. 2010 Mar;57(3):437-43. doi: 10.1016/j.eururo.2009.02.041. Epub 2009 Mar 13. PMID 19303197
- [Background] Won AC, Gurney H, Marx G, De Souza P, Patel MI. Primary treatment of the prostate improves local palliation in men who ultimately develop castrate-resistant prostate cancer. BJU Int. 2013 Aug;112(4):E250-5. doi: 10.1111/bju.12169. PMID 23879909
- [Background] Tzelepi V, Efstathiou E, Wen S, Troncoso P, Karlou M, Pettaway CA, Pisters LL, Hoang A, Logothetis CJ, Pagliaro LC. Persistent, biologically meaningful prostate cancer after 1 year of androgen ablation and docetaxel treatment. J Clin Oncol. 2011 Jun 20;29(18):2574-81. doi: 10.1200/JCO.2010.33.2999. Epub 2011 May 23. PMID 21606419
- [Background] Krupski TL, Stukenborg GJ, Moon K, Theodorescu D. The relationship of palliative transurethral resection of the prostate with disease progression in patients with prostate cancer. BJU Int. 2010 Nov;106(10):1477-83. doi: 10.1111/j.1464-410X.2010.09356.x. PMID 20977594
- [Background] Michielsen DP, Coomans D, Engels B, Braeckman JG. Bipolar versus monopolar technique for palliative transurethral prostate resection. Arch Med Sci. 2010 Oct;6(5):780-6. doi: 10.5114/aoms.2010.17095. Epub 2010 Oct 26. PMID 22419939
- [Background] Marszalek M, Ponholzer A, Rauchenwald M, Madersbacher S. Palliative transurethral resection of the prostate: functional outcome and impact on survival. BJU Int. 2007 Jan;99(1):56-9. doi: 10.1111/j.1464-410X.2006.06529.x. Epub 2006 Oct 11. PMID 17034496
- [Background] Heidenreich A, Porres D, Pfister D. The Role of Palliative Surgery in Castration-Resistant Prostate Cancer. Oncol Res Treat. 2015;38(12):670-7. doi: 10.1159/000442268. Epub 2015 Nov 23. PMID 26632812
- [Background] Brierly RD, Mostafid AH, Kontothanassis D, Thomas PJ, Fletcher MS, Harrison NW. Is transurethral resection of the prostate safe and effective in the over 80-year-old? Ann R Coll Surg Engl. 2001 Jan;83(1):50-3. PMID 11212452
- [Background] Sciarra A, Barentsz J, Bjartell A, Eastham J, Hricak H, Panebianco V, Witjes JA. Advances in magnetic resonance imaging: how they are changing the management of prostate cancer. Eur Urol. 2011 Jun;59(6):962-77. doi: 10.1016/j.eururo.2011.02.034. Epub 2011 Feb 23. PMID 21367519
- [Background] Haider MA, van der Kwast TH, Tanguay J, Evans AJ, Hashmi AT, Lockwood G, Trachtenberg J. Combined T2-weighted and diffusion-weighted MRI for localization of prostate cancer. AJR Am J Roentgenol. 2007 Aug;189(2):323-8. doi: 10.2214/AJR.07.2211. PMID 17646457
- [Background] Arora R, Koch MO, Eble JN, Ulbright TM, Li L, Cheng L. Heterogeneity of Gleason grade in multifocal adenocarcinoma of the prostate. Cancer. 2004 Jun 1;100(11):2362-6. doi: 10.1002/cncr.20243. PMID 15160339
- [Background] Karavitakis M, Winkler M, Abel P, Livni N, Beckley I, Ahmed HU. Histological characteristics of the index lesion in whole-mount radical prostatectomy specimens: implications for focal therapy. Prostate Cancer Prostatic Dis. 2011 Mar;14(1):46-52. doi: 10.1038/pcan.2010.16. Epub 2010 May 25. PMID 20498680
- [Background] Valerio M, Cerantola Y, Eggener SE, Lepor H, Polascik TJ, Villers A, Emberton M. New and Established Technology in Focal Ablation of the Prostate: A Systematic Review. Eur Urol. 2017 Jan;71(1):17-34. doi: 10.1016/j.eururo.2016.08.044. Epub 2016 Aug 29. PMID 27595377
- [Background] Mearini L, Porena M. Transrectal high-intensity focused ultrasound for the treatment of prostate cancer: past, present, and future. Indian J Urol. 2010 Jan-Mar;26(1):4-11. doi: 10.4103/0970-1591.60436. PMID 20535278
- [Background] Lafon C, Koszek L, Chesnais S, Theillere Y, Cathignol D. Feasibility of a transurethral ultrasound applicator for coagulation in prostate. Ultrasound Med Biol. 2004 Jan;30(1):113-22. doi: 10.1016/j.ultrasmedbio.2003.10.009. PMID 14962615
- [Background] Ross AB, Diederich CJ, Nau WH, Gill H, Bouley DM, Daniel B, Rieke V, Butts RK, Sommer G. Highly directional transurethral ultrasound applicators with rotational control for MRI-guided prostatic thermal therapy. Phys Med Biol. 2004 Jan 21;49(2):189-204. doi: 10.1088/0031-9155/49/2/002. PMID 15083666
- [Background] Chopra R, Baker N, Choy V, Boyes A, Tang K, Bradwell D, Bronskill MJ. MRI-compatible transurethral ultrasound system for the treatment of localized prostate cancer using rotational control. Med Phys. 2008 Apr;35(4):1346-57. doi: 10.1118/1.2841937. PMID 18491529
- [Background] Boyes A, Tang K, Yaffe M, Sugar L, Chopra R, Bronskill M. Prostate tissue analysis immediately following magnetic resonance imaging guided transurethral ultrasound thermal therapy. J Urol. 2007 Sep;178(3 Pt 1):1080-5. doi: 10.1016/j.juro.2007.05.011. Epub 2007 Jul 20. PMID 17644137
- [Background] Chopra R, Tang K, Burtnyk M, Boyes A, Sugar L, Appu S, Klotz L, Bronskill M. Analysis of the spatial and temporal accuracy of heating in the prostate gland using transurethral ultrasound therapy and active MR temperature feedback. Phys Med Biol. 2009 May 7;54(9):2615-33. doi: 10.1088/0031-9155/54/9/002. Epub 2009 Apr 8. PMID 19351975
- [Background] Burtnyk M, Chopra R, Bronskill MJ. Quantitative analysis of 3-D conformal MRI-guided transurethral ultrasound therapy of the prostate: theoretical simulations. Int J Hyperthermia. 2009 Mar;25(2):116-31. doi: 10.1080/02656730802578802. PMID 19337912
- [Background] Siddiqui K, Chopra R, Vedula S, Sugar L, Haider M, Boyes A, Musquera M, Bronskill M, Klotz L. MRI-guided transurethral ultrasound therapy of the prostate gland using real-time thermal mapping: initial studies. Urology. 2010 Dec;76(6):1506-11. doi: 10.1016/j.urology.2010.04.046. Epub 2010 Aug 14. PMID 20709381
- [Background] Partanen A, Yerram NK, Trivedi H, Dreher MR, Oila J, Hoang AN, Volkin D, Nix J, Turkbey B, Bernardo M, Haines DC, Benjamin CJ, Linehan WM, Choyke P, Wood BJ, Ehnholm GJ, Venkatesan AM, Pinto PA. Magnetic resonance imaging (MRI)-guided transurethral ultrasound therapy of the prostate: a preclinical study with radiological and pathological correlation using customised MRI-based moulds. BJU Int. 2013 Aug;112(4):508-16. doi: 10.1111/bju.12126. Epub 2013 Jun 7. PMID 23746198
- [Background] Burtnyk M, Hill T, Cadieux-Pitre H, Welch I. Magnetic resonance image guided transurethral ultrasound prostate ablation: a preclinical safety and feasibility study with 28-day followup. J Urol. 2015 May;193(5):1669-75. doi: 10.1016/j.juro.2014.11.089. Epub 2014 Nov 22. PMID 25464003
- [Background] Sammet S, Partanen A, Yousuf A, Sammet CL, Ward EV, Wardrip C, Niekrasz M, Antic T, Razmaria A, Farahani K, Sokka S, Karczmar G, Oto A. Cavernosal nerve functionality evaluation after magnetic resonance imaging-guided transurethral ultrasound treatment of the prostate. World J Radiol. 2015 Dec 28;7(12):521-30. doi: 10.4329/wjr.v7.i12.521. PMID 26753067
- [Background] Chopra R, Colquhoun A, Burtnyk M, N'djin WA, Kobelevskiy I, Boyes A, Siddiqui K, Foster H, Sugar L, Haider MA, Bronskill M, Klotz L. MR imaging-controlled transurethral ultrasound therapy for conformal treatment of prostate tissue: initial feasibility in humans. Radiology. 2012 Oct;265(1):303-13. doi: 10.1148/radiol.12112263. Epub 2012 Aug 28. PMID 22929332
- [Background] Chin JL, Billia M, Relle J, Roethke MC, Popeneciu IV, Kuru TH, Hatiboglu G, Mueller-Wolf MB, Motsch J, Romagnoli C, Kassam Z, Harle CC, Hafron J, Nandalur KR, Chronik BA, Burtnyk M, Schlemmer HP, Pahernik S. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue in Patients with Localized Prostate Cancer: A Prospective Phase 1 Clinical Trial. Eur Urol. 2016 Sep;70(3):447-55. doi: 10.1016/j.eururo.2015.12.029. Epub 2016 Jan 6. PMID 26777228
- [Background] Ramsay E, Mougenot C, Kohler M, Bronskill M, Klotz L, Haider MA, Chopra R. MR thermometry in the human prostate gland at 3.0T for transurethral ultrasound therapy. J Magn Reson Imaging. 2013 Dec;38(6):1564-71. doi: 10.1002/jmri.24063. Epub 2013 Feb 25. PMID 23440850
- [Background] Ramsay E, Mougenot C, Staruch R, Boyes A, Kazem M, Bronskill M, Foster H, Sugar L, Haider M, Klotz L, Chopra R. Evaluation of Focal Ablation of Magnetic Resonance Imaging Defined Prostate Cancer Using Magnetic Resonance Imaging Controlled Transurethral Ultrasound Therapy with Prostatectomy as the Reference Standard. J Urol. 2017 Jan;197(1):255-261. doi: 10.1016/j.juro.2016.06.100. Epub 2016 Aug 18. PMID 27545572
- [Background] Sommer G, Pauly KB, Holbrook A, Plata J, Daniel B, Bouley D, Gill H, Prakash P, Salgaonkar V, Jones P, Diederich C. Applicators for magnetic resonance-guided ultrasonic ablation of benign prostatic hyperplasia. Invest Radiol. 2013 Jun;48(6):387-94. doi: 10.1097/RLI.0b013e31827fe91e. PMID 23462673
- [Background] Roach M 3rd, Hanks G, Thames H Jr, Schellhammer P, Shipley WU, Sokol GH, Sandler H. Defining biochemical failure following radiotherapy with or without hormonal therapy in men with clinically localized prostate cancer: recommendations of the RTOG-ASTRO Phoenix Consensus Conference. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):965-74. doi: 10.1016/j.ijrobp.2006.04.029. PMID 16798415
- [Derived] Wright C, Makela P, Bigot A, Anttinen M, Bostrom PJ, Blanco Sequeiros R. Deep learning prediction of non-perfused volume without contrast agents during prostate ablation therapy. Biomed Eng Lett. 2022 Nov 8;13(1):31-40. doi: 10.1007/s13534-022-00250-y. eCollection 2023 Feb. PMID 36711157
- [Derived] Anttinen M, Makela P, Nurminen P, Yli-Pietila E, Suomi V, Sainio T, Saunavaara J, Taimen P, Blanco Sequeiros R, Bostrom PJ. Palliative MRI-guided transurethral ultrasound ablation for symptomatic locally advanced prostate cancer. Scand J Urol. 2020 Dec;54(6):481-486. doi: 10.1080/21681805.2020.1814857. Epub 2020 Sep 8. PMID 32897169
- [Derived] Anttinen M, Yli-Pietila E, Suomi V, Makela P, Sainio T, Saunavaara J, Eklund L, Blanco Sequeiros R, Taimen P, Bostrom PJ. Histopathological evaluation of prostate specimens after thermal ablation may be confounded by the presence of thermally-fixed cells. Int J Hyperthermia. 2019;36(1):915-925. doi: 10.1080/02656736.2019.1652773. PMID 31466481